CLINICAL TRIAL: NCT02577601
Title: Determining the Impact of Combined Hormonal Contraceptives on Ulipristal Acetate
Brief Title: Impact of Combined Hormonal Contraceptives on UPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Alison Edelman, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OHSU IRB 11784
Record Dates: First submitted 2015-08-05; First posted 2015-10-16 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Contraception
Keywords: Emergency contraception; Birth Control Pills
MeSH Terms: interventions — ulipristal acetate; Levonorgestrel; Ethinyl Estradiol-Norgestrel Combination; Drugs, Generic; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UPA Only (Active Comparator): During the first treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10). Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier.
  Interventions: Drug: Ulipristal Acetate
- Washout Cycle (No Intervention): The month following this first treatment month (washout-cycle),there will be no study visits during this menstrual cycle but there will be contact with study staff (1 or 2 times) by telephone or email to discuss any health changes that are experiencing.
- UPA + COC (Active Comparator): During the second treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10) and then 2 days later start birth control pills. Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier.
  Interventions: Drug: Ulipristal Acetate; Drug: Levonorgestrel (LNG)/Ethinyl estradiol birth control pill

INTERVENTIONS:
Drug: Ulipristal Acetate
  Other Names: UPA; Ella
  Arms: UPA + COC; UPA Only
Drug: Levonorgestrel (LNG)/Ethinyl estradiol birth control pill
  Other Names: portia (generic); birth control pills
  Arms: UPA + COC

SUMMARY:
The purpose of this research study is to determine if taking a birth control pill effects how well an emergency contraceptive pill called Ulipristal acetate (UPA) works. This type of emergency contraceptive is the most effective oral method available. However, this medication is an anti-progestin and most regular forms of birth control contain progestin (a female hormone). It is unknown if taking the two close together may make the emergency contraceptive not work well. The overall goal of this research is to improve the effectiveness of contraception for women and to better counsel women.

DETAILED DESCRIPTION:
Emergency contraception (EC) provides women with an additional line of defense against unintended pregnancy during an act of unprotected intercourse. An antiprogestin, ulipristal acetate (UPA; ellaTM), has emerged as one of the most effective oral options. However, there is currently a lack of information regarding the practical use of UPA. Basic science studies have shown that UPA binds to and prevents progesterone receptor from working, leading to the possible concern that hormonal contraceptives, like the birth control pill, would prevent UPA from working. Ideally, women should start their regular method of birth control soon after EC use but by doing this, they may prevent the UPA EC from working. A woman could just delay starting her regular method of birth control but then she is still at risk for pregnancy.

This proposal has been designed to address this gap in knowledge and will focus on the impact of the birth control pill on UPA's ability to delay ovulation (or the release of an egg). Subjects will undergo a referent cycle UPA only (Cycle 1, 1 month), followed by a washout cycle (Cycle 2, 1 month) and finally UPA with combined oral contraceptives (COCs) dosed 2 days later (Cycle 3, 1 month treatment cycle). The hypothesis is that starting the birth control pill shortly after UPA adversely impacts UPA's ability to delay ovulation.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women aged 18 to 35 with regular menses (every 21-35 days).
* Normal BMI
* Proven ovulation with a screening serum progesterone of >3ng/mL
* Willing to use condoms (if sexually active with a male partner), willing to not have sex with men during the study, or have had a tubal ligation (or have a partner who has had a vasectomy) or have a copper intrauterine device (IUD).

Exclusion Criteria:

* Known intolerance or allergy to any of the study medication
* Known metabolic disorders including polycystic ovarian syndrome or uncontrolled thyroid disorder
* Overweight or obese BMI
* Any Centers for Disease Control and Prevention (CDC) Medical eligibility criteria category 3 or 4 for combined oral contraception (COC) use 12.
* Pregnancy, breastfeeding, or seeking pregnancy; recent (8 week) use of hormonal contraception
* Current use of drugs that interfere with metabolism of sex steroids
* Smokers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
PI acknowledges willingness to share data and materials with other investigators through established means. Data will be presented via presentation and publication. Transfer of resources is subject to the acceptance of a Materials Transfer Agreement as required by policy at Oregon Health & Science University (OHSU). OHSU complies with NIH policy on Sharing Research Data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Cycles: UPA only: During the first treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10). Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier. Cycle 1: Ulipristal Acetate
  UPA+COC: During the second treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10) and then 2 days later start birth control pills. Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier. Cycle 3: Ulipristal Acetate and Levonorgestrel (LNG)/Ethinyl estradiol birth control pill
Period: UPA Only (1 Month)
Arm/Group | Treatment Cycles
Started | 36
Completed | 36
Not Completed | 0
Period: Washout (1 Month)
Arm/Group | Treatment Cycles
Started | 33
Completed | 33
Not Completed | 0
Period: UPA+COC (1 Month)
Arm/Group | Treatment Cycles
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Cycles: During the first treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10). Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier. Cycle 1: Ulipristal Acetate
  The month following this first treatment month (washout-cycle),there will be no study visits during this menstrual cycle but there will be contact with study staff (1 or 2 times) by telephone or email to discuss any health changes that are experiencing.
  During the second treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10) and then 2 days later start birth control pills. Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier. Cycle 3: Ulipristal Acetate and Levonorgestrel (LNG)/Ethinyl estradiol birth control pill
Arm/Group | All Cycles
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Follicle Rupture
Description: Following dosing with UPA, subjects underwent daily visits with ultrasound monitoring until evidence of follicle rupture (complete disappearance or >50% reduction of the mean size of the leading follicle).
Time Frame: within 5 days of taking the study drug
Measure: Count of Participants; unit: Participants
Groups:
- UPA Only: During the first treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10). Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier.
  Ulipristal Acetate
- UPA + COC: During the second treatment month, 1 dose of the study medication ulipristal acetate (UPA) will be given when the follicle is a certain size (approximately cycle day 10) and then 2 days later start birth control pills. Following this, there will be daily study visits for 7 days unless evidence of ovulation occurs earlier.
  Ulipristal Acetate
  Levonorgestrel (LNG)/Ethinyl estradiol birth control pill
Arm/Group | UPA Only | UPA + COC
Number analyzed (Participants) | 33 | 33
Participants | 1 | 9

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | UPA Only | Washout Cycle | UPA + COC
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 1/36 | 0/33 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UPA Only (N=36) | Washout Cycle (N=33) | UPA + COC (N=33)
Malar rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — One subject reported a significant malar rash several hours after UPA dosing in Cycle 1 that resolved on its own and did not reoccur with UPA dosing in Cycle 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02577601/Prot_SAP_000.pdf